CLINICAL TRIAL: NCT00188812
Title: Open-Label, Multicentre, One Year Extension of the Evaluation of the Safety of Donepezil Hcl in Patients With Dementia Associated With Cerebrovascular Disease
Brief Title: Safety of Donepezil in Patients With Dementia Associated With Cerebrovascular Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-0725-AE; E2020-A001-320
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2005-09

CONDITIONS: Dementia Associated With Cerebrovascular Disease
Keywords: dementia; stroke
MeSH Terms: conditions — Dementia; Stroke | interventions — Donepezil

INTERVENTIONS:
Drug: donepezil hcl

SUMMARY:
one year extension study following a previous double-blind study to evaluate safety of the drug

DETAILED DESCRIPTION:
A one year extension study for patients who completed E2020-A001-319. Patients will receive 5my donepezil daily for the first 8 weeks and will be assessed by the incidence of advere events, changes in physical exams, ECG and clinical lab determinations. The results will be assessed 6 timues during the year. After 8 week, the investigator may increase the dose to 10mg/day if the patient if the patients show satisfactory tolerability. Six psychometric scales will also be evaluatd.

ELIGIBILITY:
Inclusion Criteria:

* must have completed previous study E2020-A001-319

Exclusion Criteria:

* absence of a reliable caregiver
* clinically significant medical condition
* recent TIA

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-05; Study Completion 2005-08

PRIMARY OUTCOMES:
safety assessments

CONTACTS AND LOCATIONS:
Overall Officials: Karl Farcnik, MD FRCP(C), Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hopital, Toronto, Ontario, Canada